CLINICAL TRIAL: NCT04052061
Title: Open-Label, Phase 1 Study of CD19 t-haNK In Subjects With Diffuse Large B-Cell Lymphoma Who Have Received 2 Or More Lines of Therapy And Are Ineligible For Transplant
Brief Title: QUILT-3.061: CD19 t-haNK in Subjects With Diffuse Large B-Cell Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial not initiated
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.061
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2022-05

CONDITIONS: Diffuse Large B Cell Lymphoma; Large-cell Lymphoma; Lymphoma, B-Cell; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, B-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CD19 t-haNK (Experimental): CD19 t-haNK will be administered to patients with Diffuse Large B-Cell Lymphoma who have received 2 or more lines of therapy and are ineligible for transplant.
  Interventions: Biological: CD19 t-haNK

INTERVENTIONS:
Biological: CD19 t-haNK — CD19 t-haNK Suspension for Infusion

SUMMARY:
Phase 1 study to assess the safety, preliminary efficacy of CD19 t-haNK and to determine the maximal tolerated dose and designate the recommended phase 2 dose in subjects with diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
Phase 1 study to assess the safety, preliminary efficacy of CD19 t-haNK and to determine the maximal tolerated dose and designate the recommended phase 2 dose in subjects with diffuse large B-cell lymphoma (DLBCL). The study will be conducted in 2 parts: part 1 will involve dose escalation and part 2 will involve expansion of the recommended phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant Institutional Review Board (IRB) or Independent Ethics Committee (IEC) guidelines.
3. Have histologically confirmed DLBCL that is refractory or relapsed after at least 2 lines of previous therapy.
4. Are ineligible for autologous stem cell transplant, allogeneic stem cell transplant or CAR T cell therapy under 1 of the following conditions:

   1. Have chemotherapy refractory disease after 2 lines of salvage chemotherapy.
   2. Have met eligibility for CAR T-cell therapy or transplant, but have refused therapy.
5. Have disease progression or relapse within 12 months after autologous or allogeneic stem cell transplant or have relapsed following CAR T-cell therapy and meet the following criteria:

   1. Had a partial response (PR) or stable disease (SD) at the 3-month disease assessment and then subsequently progressed > 3 months after first CAR T-cell therapy.
   2. Have confirmed CD19 tumor expression by biopsy after disease progression and prior to retreatment.
   3. Have not received subsequent therapy for the treatment of lymphoma post CAR T-cell therapy.
   4. Toxicities related to conditioning chemotherapy (fludarabine and cyclophosphamide), with the exception of alopecia, have resolved to ≤ grade 1 or returned to baseline prior to retreatment.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Have at least 1 measurable lesion and/or non-measurable disease evaluable in accordance with RECIST Version 1.1.
8. Must have a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen obtained following the conclusion of the most recent anticancer treatment and be willing to release the specimen for exploratory tumor molecular profiling. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
9. Must be willing to provide pre- and post-infusion blood samples for exploratory analyses.
10. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
11. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception while on study and for at least 5 months after the last dose of CD19 t-haNK for Infusion. Non-sterile male subjects must agree to use a condom while on study and for up to 5 months after the last dose of CD19 t-haNK for Infusion. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. Body weight at screening of ≤ 50 kg.
2. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
3. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
4. History of organ transplant requiring immunosuppression.
5. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
6. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count (ANC) < 750 cells/mm3.
   2. Platelet count < 75,000 cells/mm3.
   3. Hemoglobin < 9 g/dL.
   4. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   5. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   6. Alkaline phosphatase (ALP) levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177

   Each study site should use its institutional ULN to determine eligibility.
7. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for human immunodeficiency virus (HIV).
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Participation in an investigational drug study or history of receiving any investigational treatment within 14 days prior to dosing for this study, except for testosterone-lowering therapy in men with prostate cancer.
13. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
14. Concurrent participation in any interventional clinical trial.
15. Pregnant and nursing women. A negative serum pregnancy test during screening and a negative pregnancy test within 72 hours prior to the first dose must be documented before CD19 t haNK for Infusion is administered to a female subject of child-bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-16 (Estimated); Primary Completion 2021-09-18 (Estimated); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
MTD or HTD and RP2D. | 1 year
  Maximum tolerated dose or highest tested dose and recommended phase 2 dose.
Incidence of DLTs and treatment-emergent adverse events | 1 year
  Incidence of DLTs and treatment-emergent adverse events (AEs) and serious AEs (SAEs), graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Clinically significant changes | 1 year
  Clinically significant changes in safety laboratory tests, physical examinations, electrocardiograms (ECGs), and vital signs, as determined by the physician and/or lab ranges.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
  ORR in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 and modified RECIST guidelines for immunotherapy trials (iRECIST).
Progression-free Survival (PFS) | 1 year
  Progression-free Survival (PFS) by RECIST Version 1.1 and iRECIST.
Overall Survival (OS) | 1 year
  OS will be evaluated using Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: No